CLINICAL TRIAL: NCT04400604
Title: Evaluation of the Natural History of Alcoholic Liver Disease According to Baseline Severity
Brief Title: Study of Alcohol-related Liver Disease in Europe
Acronym: SALVE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_04; 2020-A00527-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-14; First posted 2020-05-22 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a genetic sample (DNA, 1 EDTA tube) serum sample (2 dry 7 ml tubes) plasma (2 heparin 7 ml tubes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: Patients with minimal risk of extensive fibrosis: TE < 5.8kPa; rule out cut-off value)
- 2: Patients with intermediate risk of fibrosis
- Patients with high risk of extensive fibrosis
- Patients with compensated cirrhosis biopsy-proven
- Patients with a first decompensation: patients with a first decompensation event of cirrhosis after exclusion of HCC.

SUMMARY:
Alcohol-induced liver injury is made up of fatty liver, fibrosis and alcoholic hepatitis (AH), elementary lesions that may occur separately, simultaneously or sequentially in a same patient. Among these histological features, alcoholic hepatitis, a necro-inflammatory process is associated with the fastest fibrosis progression leading to cirrhosis in 40% of cases and a pivotal lesion driving increased risk of liver decompensation.

The non-invasive methods for the diagnosis of fibrosis open new perspectives for a better understanding of the natural history of disease-progression from early injury to the cirrhotic stage, for the identification of subgroup patients at risk of developing cirrhosis at medium term and for proposing a strategy of screening of patients with extensive cirrhosis at risk of liver-threatening events. There is an urgent need to perform studies in asymptomatic heavy drinkers in order to identify cut-offs associated with significant risk of development of cirrhosis at medium term. Such objectives require large-scale screening of heavy drinkers. Each of non-invasive methods have been tested to predict with of extensive fibrosis with a high predictive performance as shown below.

A screening policy cannot be accepted without answering the following questions: a) are the requirements of public health screening fulfilled? b) Is the group of patients undergoing screening defined? c) is there a reliable method for of testing? Indeed, the detection of a disease is subject to certain public health requirements and may be proposed to health authorities only if it modifies the management of subjects screened. In the specific case of mass screening of liver fibrosis in heavy drinkers, only the detection of extensive fibrosis could fulfill this criterion because of the potential survival benefit resulting from the screening of hepatocellular carcinoma (HCC) in patients with extensive fibrosis. Indeed, recent studies have found that the probability of receiving curative treatment of HCC was significantly higher in patients who received a six-month surveillance ultrasound. Therefore, the detection of extensive fibrosis seems reasonable in the light of these studies when considering that the yearly risk of development of HCC in the subgroup of heavy drinkers with extensive fibrosis is approximately 3%.

Taking into account the above scientific arguments, the most recent EASL clinical practical guidelines on ALD recommend longitudinal studies using non-invasive tools to evaluate screening of extensive fibrosis and disease progression in heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Active alcohol excessive consumption defined as > 210 g per week for men and> 140 g per week for women during the previous year.
* Patients with high risk of alcoholic-related liver disease can be included only if the following assessment were available: Abdominal Ultrasound / Ultrasound elastography pulse (FibroScan®) / FibroTest®, AshTest® and LCR1-LCR2® (cost will be supported by Biopredictive) / Non-patented methods: Forns Index; Fib-4, Hepascore®/ Absolute values should be provided for all these methods.

For patient in whom liver stiffness measurements were uninterpretable (unavailable results) only those with FibroTest® and LCR1 and LCR2 measurements can be included.

Results of FibroScan® were considered unavailable based on following criteria: When no value was obtained after at least 10 shots (valid shot=0) OR If SR (Success Rate), the ratio of valid shots to the total number of shots at least 60% OR IQR (InterQuartil Range reflecting variability of measurements) less than 30% of the median LSM (Liver Stiffness Measure) value (IQR≤LSM≤30%).

* Patients must provide written informed consent and agree to have blood stored for the study and tissue stored for those in whom physicians performed liver biopsy according their clinical practice.
* Patients should agree to participate for at least 5-year follow-up.
* Patients with social insurance

Exclusion Criteria:

For all study groups, the following exclusion criteria will be applied:

* Evidence of other forms of known chronic liver disease including:Positive test result at baseline for hepatitis B surface antigen or positive serology of hepatitis C virus infection (regardless PCR results)/ Autoimmune liver disease / Known or suspected HCC
* Any previous episode of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding before current hospitalization and/or inclusion in the study
* Known positivity for human immunodeficiency virus infection.
* Terminal extrahepatic illness defined as: All conditions evolved into a clinical stage to limit the patient's functional status (e.g.: heart failure, renal failure, neurological or respiratory diseases, or any other disabling diseases etc. …).
* Other medical conditions that may diminish life expectancy to <2 years.
* Known extra-hepatic cancers with the exception of basal cell skin cancer.
* Any other condition that, in the opinion of the Investigator, would impede completion of the study (eg: Homeless, non-compliant patients…).
* Mental instability or incompetence, such that the validity of informed consent is uncertain.
* Lack of informed consent or refusal to participate for follow up evaluation.
* A condition in which repeated blood draws pose more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access.
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in adults patients with active alcohol excessive consumption defined as > 210 g per week for men and> 140 g per week for women during the previous year.
  Patients with high risk of alcoholic-related liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
A first occurrence of clinical diagnosis of cirrhosis and/or its complications(for patients of group 1 and 2) | at five years
  The primary endpoint is a composite criterion defined as a first occurrence of clinical diagnosis of cirrhosis and/or its complications.
  The primary endpoint will be held in the presence of any of the following criteria:
  Clinical cirrhosis Or Hepatocellular carcinoma (HCC) Or Histological diagnosis of cirrhosis on liver biopsy Or Biological features of liver dysfunction: INR≥1.5 in the presence of one of the following features: platelet count <100 000, albumin <35g, bilirubin > 2* ULN it will assess the risk of clinical diagnosis of cirrhosis and/or its complications in heavy drinkers classified according to non-invasive methods at minimal or intermediate risk of extensive fibrosis (groups 1,2).

SECONDARY OUTCOMES:
cumulative incidence of cirrhosis and/or complications by treating death as competing risk.(for patients of group 3) | at five years
  measure the risk of clinical diagnosis of cirrhosis and/or its complications in heavy drinkers classified according to non-invasive methods at high risk of extensive fibrosis (group 3).
All-cause of death | at five years
  all-cause mortality in groups of heavy drinkers (Groups 1,2,3) and cirrhotic groups (Groups 4 et 5)
Biobanking of liver tissue and blood samples for further analyses such as cirrhosis disease studies | at five years
  A multi-national registry of liver tissue and blood samples (bio-bank collection) to get more insights in risk of development of cirrhosis and disease-progression of cirrhosis
LCR1/LCR2 test | at five years
  Measure the performance of LCR1 and LCR2 to predict risk of development of hepatocellular carcinoma (All Groups) LCR1 test combines (using Cox model) hepatoprotective proteins (apolipoproteinA1, haptoglobin) with known risk factors (gender, age, gamma-glutamyltranspeptidase), and a marker of fibrosis (alpha2-macroglobulin). To increase the specificity, the LCR2 test was developed by combining the components of LCR1 to alpha-fetoprotein. The predetermined cutoffs are <0.015 for low-LCR1, and <0.044 for low-LCR2 will be tested as the rule-out values to exclude a risk of hepatocellular carcinoma.
Brief Drinking Questionnaire (Audit-C) | at five years
  The AUDIT-C (Alcohol Use Disorder Identification Test) quantifies alcohol misuse, based on 3 questions posed to patients about their consumption habits. It was adapted from the first three questions of the AUDIT.
  The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). Each question has 5 answer choice.
  In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Alcohol consumption according to the WHO category | at five years
  Patterns of alcohol consumption will be classified according the 5 risks levels (Abstinence, Low risk, Medium risk, high risk, very high risk).
The occurrence of decompensation of cirrhosis | at five years
  To determine the 5-year risk of first decompensation in patients with biopsy-proven compensated cirrhosis at inclusion (Group 4)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mathurin, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No